CLINICAL TRIAL: NCT02005679
Title: Transposition of the Mini-Mental State in Sign Language
Brief Title: Mini-Mental State (MMS-LS) and Sign Language
Acronym: MMS-LS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0008
Record Dates: First submitted 2013-11-22; First posted 2013-12-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prelingual Deafness; Retention Disorders, Cognitive
Keywords: Prelingual Deafness; Retention Disorders, Cognitive; Sign language; Mini-Mental State
MeSH Terms: conditions — Deafness; Memory Disorders; Sign Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- deaf persons with potential dementia (Experimental)
  Interventions: Behavioral: application of the mini-mental state test

INTERVENTIONS:
Behavioral: application of the mini-mental state test

SUMMARY:
In France the prevalence of pre-lingual deafness is between 1 and 1.4 per 1000 habitants, and according to very conservative estimates, about 44 000 deaf persons use the sign language. Additionally, the prevalence of dementia in France is close to 1% (850 000 dements for a total population of 65 millions). The prevalence of dementia in pre-lingual deaf adults has also been described and is between 1 and 1.4 /100 000 habitants.

The Mini Mental State Examination (MMSE) of Folstein is a test recommended to perform the cognitive evaluation for the detection of mental disorders including dementia, and a consensual French version exists prepared by GRECO (Group of Research and Cognitive Assessments). However, to date, there are no simple, rapid and validated screening tests to study cognitive disorders in deaf persons who use the sign language. The only tests available allow a late diagnosis avoiding an optimal treatment of the patients.

DETAILED DESCRIPTION:
The objective of this study is to assess the intrinsic quality of the tool MMS-LS, a mini-mental state examination that has been adapted to the sign language in order to monitor cognitive disorders in deaf people who speak sign language.

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years
* Pre-lingual deafness
* Use of French sign language

Exclusion Criteria:

* Refusal to sign the consent
* Severe visual impairment with lower acuity (less than 0.5)
* Severe motor difficulties impeding the practice of sign language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Assessment of internal consistency of MMS-LS test for the diagnosis of cognitive impairment among deaf patients by a correlation analysis followed by Cronbach's alpha test | At baseline, 1 year and 2 years follow-up visits

SECONDARY OUTCOMES:
Description of MMS-LS test results | Baseline
  Explanatory Factors are: age, education level, characteristics of the sign language(fluency level, learning age, usage frequency, usage by other family members)
Diagnostic performance and predictive values of MMS-LS test for acquired dementia. | Baseline, 1 year and 2 years follow-up visits
  Sensitivity, specificity, positive and negative predictive values.
Correlation between MMS-LS score and CDR level | Baseline, 1 year and 2 years follow-up visits
  We also check that patients having a suspicious CDR (0.5) have a superior MMS-LS score compared to patients having a CDR ≥ 1.
Diagnostic performance and predictive values of MMS-LS test for suspected dementia. | Baseline, 1 year and 2 years follow-up visits
  Sensitivity, specificity, positive and negative predictive values

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Drion, MD, Study Director — Groupement des Hôpitaux de l'Institut Catholique de Lille, Unité d'Accueil et de Soins des Sourds en Langue des Signes et Réseau Sourds et Santé; Amélie Lansiaux, MD, Study Chair — Groupement des Hôpitaux de l'Institut Catholique de Lille, Medical Research Department; Isabelle Ridoux, MD, Principal Investigator — CHU de Rennes, Hôpital de Pontchaillou; Corine Gilda Scemama-Ammar, MD, Principal Investigator — Hôpital de la Conception, Pôle psychiatrie, Marseille; Charlotte Crinquette, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille; Isabelle Bouillevaux, MD, Principal Investigator — CHRU de Nancy, Unité Régionale d'Accueil et de Soins pour Sourds et malentendants
Locations (4):
- France (4):
  - Hôpital de la Conception, Pôle psychiatrie Centre, Marseille, Bouches-du-Rhône
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, Hauts-de-France
  - CHU de Rennes, Hôpital de Pontchaillou, Rennes, Ille-et-Vilaine
  - Unité Régionale d'Accueil et de Soins pour Sourds et malentendants - CHRU Nancy, Nancy, Meurthe-et-Moselle